CLINICAL TRIAL: NCT02137889
Title: A Phase 1, Muticenter, Open-label, Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VAY736 When Administered Intravenously in Relapsed or Refractory Chronic Lymphocytic Leukemia Patients
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VAY736 in Relapsed or Refractory CLL Patients
Acronym: VAY736Y
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated on 04Oct2013 for business reasons after being on hold for 10 months. Early termination was not due to safety concerns.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAY736Y2101; 2011-005485-38 (EudraCT Number)
Record Dates: First submitted 2014-04-29; First posted 2014-05-14 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL)
Keywords: CLL
MeSH Terms: conditions — Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ianalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1- relapsed/refractory CLL patients (Experimental): Patients with relapsed/refractory CLL with two or three prior treatment regimens
  Interventions: Drug: VAY736
- Arm 2 - rituximab or ofatumumab refractory CLL patients (Experimental): Patients with relapsed/refractory CLL with four or more prior treatment regimens
  Interventions: Drug: VAY736

INTERVENTIONS:
Drug: VAY736 — VAY736 is a human immunoglobulin of the G class (IgG1/k) monoclonal antibody (mAb) designed to specifically bind the BAFF receptor. VAY736 binds primarily to B-cells through its fragment antigen binding (Fab) region, in human whole blood and spleen samples; it does not bind to natural killer (NK) cells, monocytes, dendritic cells, granulocytes, or platelets.

SUMMARY:
This study will assess the safety and preliminary efficacy of escalating doses of VAY736 in relapsed or refractory CLL patients.

DETAILED DESCRIPTION:
This Phase 1, multicenter, open-label, study will investigate the safety, pharmacokinetics, pharmacodynamics, and preliminary antil-CLL activity of VAY736 in patients with relapsed/refractory CLL who have received at least two prior regimens. The study will include one arm in the dose escalation phase and two arms in the dose expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Dose escalation: Relapsed/refractory CLL following at least -two prior treatment regimen
* Dose expansion:

  * Arm 1: Relapsed/refractory CLL following two to three prior treatment regimens
  * Arm 2: Relapsed/refractory CLL following four or more prior treatment regimens
* Discontinued any previous anti-cancer and investigational therapy including radiation, radioimmunotherapy, and monoclonal antibody therapy for at least 28 days or 5 half-lives of the investigational product, whichever is longer, before study treatment administration, and must have recovered fully from the adverse effects of such treatment before beginning study treatment
* Discontinued prior alemtuzumab therapy for at least 6 months
* Age 18 years
* Eastern cooperative oncology group (ECOG) performance status grade ≤ 1
* Life expectancy > 3 months
* Meet the following laboratory criteria (must be obtained within 14 days of enrollment):

  • Adequate end-organ function as assessed by laboratory tests, as specified in the protocol.
* Written informed consent obtained prior to any screening procedures

Exclusion Criteria:

* Major surgery within 28 days before study treatment or have not recovered fully from the adverse effects of any major or minor surgical procedures before study treatment
* History of another primary malignancy that is currently clinically significant or currently requires active intervention (except adequately treated in situ carcinoma of the cervix or non-melanoma carcinoma of the skin or any other curatively treated malignancy that has not been treated in the prior 3 months or expected to require treatment for recurrence during the course of the study).
* Prior anaphylactic or other severe infusion reaction such that the patient is unable to tolerate human immunoglobulin or monoclonal antibody administration
* Clinically significant central nervous system disease
* Myocardial infarction within 6 months prior to enrollment or New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or significant conduction system abnormalities in the opinion of the investigator
* History of an active infection requiring systemic therapy within 14 days before study treatment. Prophylactic antibiotics and antiviral therapies are permitted.
* Active autoimmune disease requiring immunosuppressive therapy
* Known history of human immunodeficiency virus (HIV) or active infection with hepatitis C virus or hepatitis B virus or any active bacterial, viral, or fungal infection requiring systemic therapy
* Ongoing corticosteroid use (>10 mg/day prednisone or equivalent)
* Pregnant or nursing (lactating) women.
* Sexually active males must use a condom during intercourse while taking the drug and for 3 months after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | 8 months
  Frequency and characteristics of DLTs. Determination of the maximum tolerated dose (MTD) and/or the recommended dose for expansion (RDE) of VAY736 when administered weekly in patients with relapsed or refractory chronic lymphocytic leukemia (CLL) (dose escalation only).

SECONDARY OUTCOMES:
Overall response rate (ORR) | 1 year
  Determine the preliminary anti-CLL (chronic lymphocytic leukemia) activity of VAY736 at the MTD/RDE in patients with relapsed or refractory CLL.
VAY736 plasma concentrations | 1 year
  Plasma concentrations to characterize the pharmaconinetics of VAY736
Blood Serum concentrations of antibodies to VAY736 | 1 year
  To assess the immunogenicity of VAY736.
Hematology parameters of VAY736 | 1 year
  To assess the pharmacodynamics of VAY736.
Number of patients with Advers Events (AEs) as a measure of safety and tolerability. | 1 year
  To assess the safety and tolerability of VAY736 by type, frequency, and severity of AEs, changes in hematology and blood chemistry values, assessments of physical examinations, vital signs, and electrocardiograms.
PharmacoKinetics (PK) parameters of VAY736 | 1 year
  PK parameters include AUC0-tlast, Cmax, T1/2
Receptor occupancy for VAY736 | 1 year
  To assess the pharmacodynamic effect of VAY736.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- H. Lee Moffitt Cancer Center & Research Institute Moffitt Cancer SC, Tampa, Florida, United States
- Novartis Investigative Site, Barcelona, Catalonia, Spain